CLINICAL TRIAL: NCT04908462
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Single and Multiple Ascending Dose in Healthy Volunteers and Autosomal Dominant Polycystic Kidney Disease Subjects Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Oral AL01211
Brief Title: To Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Oral AL01211 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AceLink Therapeutics, Inc. (Industry)
Collaborators: Novotech (Australia) Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: AL01211-101
Record Dates: First submitted 2021-05-18; First posted 2021-06-01 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Autosomal Dominant Polycystic Kidney
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part A Healthy volunteers: Single ascending doses (Experimental)
  Interventions: Drug: AL01211 or Placebo (Part A)
- Part B Healthy Volunteers Multiple ascending doses (Experimental)
  Interventions: Drug: AL01211 or Placebo (Part B)

INTERVENTIONS:
Drug: AL01211 or Placebo (Part A) — Five dose groups with doses ranging from 2mg to 60 mg
  Arms: Part A Healthy volunteers: Single ascending doses
Drug: AL01211 or Placebo (Part B) — Five dose groups with doses ranging from 2-60 mg daily. Each separate dose given for 14 days
  Arms: Part B Healthy Volunteers Multiple ascending doses

SUMMARY:
The study is designed to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of Oral AL01211 in healthy volunteers

DETAILED DESCRIPTION:
This study is a Phase 1, first in human (FIH), randomized, double-blind, placebo-controlled study of AL01211 in healthy adult participants

The study consists of two parts:

Part A will investigate the safety, tolerability, pharmacokinetics, and pharmacodynamics of AL01211 in a single ascending dose escalation study in approximately 40 healthy adult participants.

Part B will investigate the safety and tolerability, pharmacokinetics, and pharmacodynamics of AL01211 in a multiple ascending dose escalation study in approximately 40 healthy adult volunteers.

ELIGIBILITY:
Inclusion Criteria:

For Part A (SAD) and Part B (MAD)

To be eligible for the study, participants must meet all of the following inclusion criteria:

1. Healthy male or female volunteers, between 18 and 55 years of age
2. Participants in good health as determined by medical history, physical examination, vital signs, ECG, and clinical laboratory tests.
3. Body Mass Index (BMI) between 20.0 and 34.9 kg/m2 (inclusive).
4. Participants who smoke no more than 2 cigarettes per day or equivalent per week (includes e-cigarettes) can be included in the study but must be willing to abstain from smoking during confinement periods.
5. Participants must have no relevant dietary restrictions,
6. Females must be non-pregnant and non-lactating, and must use an acceptable, highly effective double contraception from Screening until at least 30 days have passed since study drug administration , including the follow-up period. Double contraception is defined as a condom AND one other form of the following:

   * Established hormonal contraception (oral contraceptive pills [OCPs], long-acting implantable hormones, and injectable hormones) for at least 1 month prior to Screening
   * A vaginal ring or an intrauterine device [IUD]
   * Documented evidence of surgical sterilization at least 6 months prior to Screening (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy, or bilateral oophorectomy) for women or vasectomy at least 90 days prior to Screening for men (with appropriate post-vasectomy documentation of the absence of sperm in semen), provided the male partner is a sole partner.
   * Women not of childbearing potential must be postmenopausal for ≥ 12 months. Postmenopausal status will be confirmed through testing of follicle-stimulating hormone (FSH) levels ≥ 40 IU/mL at Screening for amenorrhoeic female participants. Females who are abstinent from heterosexual intercourse will also be eligible.

   Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not considered highly effective methods of birth control. Participant complete abstinence for the duration of the study and for 1 month after the last study treatment is acceptable.

   Female participants who exclusively are in same sex relationships are not required to use contraception.

   - Males must be surgically sterile (> 90 days since vasectomy with no viable sperm), abstinent, or if engaged in sexual relations with a woman of childbearing potential (WOCBP), the participant and his partner must be surgically sterile (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy, bilateral oophorectomy) or using an acceptable, highly effective contraceptive method from Screening until at least 90 days have passed since study drug administration, including the follow-up period. Acceptable methods of contraception include the use of condoms and the use of an effective contraceptive for the female partner that includes: OCPs, long-acting implantable hormones, injectable hormones, a vaginal ring, or an IUD. Participants with same sex partners (abstinence from penile-vaginal intercourse) are eligible when this is their preferred and usual lifestyle.

   WOCBP must have a negative pregnancy test at Screening and Day -1 and be willing to have additional pregnancy tests as required throughout the study.

   Males must not donate sperm for at least 90 days after the last dose of AL01211.
7. Participants must have the ability and willingness to attend the necessary visits to the CRU.
8. Must sign an informed consent form (ICF) indicating that they understand the purpose of, and procedures required for the study and are willing to participate in the study.

Exclusion Criteria:

For Part A (SAD) and Part B (MAD)

A participant who meets any of the following exclusion criteria must be excluded from the study:

1. Any concomitant disease, condition, or treatment that could interfere with the conduct of the study,.
2. History or symptoms of significant psychiatric disease,
3. History or evidence of significant hepatic or renal disease or impairment, including clinically significant abnormalities in laboratory test results (including complete blood count, chemistry panel including kidney panel and liver function tests, and urinalysis).
4. Evidence of an active or suspected cancer or a history of malignancy for at least 5 years, except for: nonmelanoma skin cancer considered cured, curatively treated localized prostate cancer, or other in situ cancer.
5. Known hypersensitivity or allergy to AL01211 or excipient contained in the drug formulation.
6. Uncontrolled hypertension of > 140/90 mm Hg despite optimal therapy.
7. Any of the following abnormal ECG findings at Screening:

   * PR interval > 210 ms or < 120 ms
   * QRS interval > 120 ms
   * QTcF interval > 450 ms
   * ST segment elevation or depression considered to be clinically significant
8. Any hepatic laboratory abnormality > 1.5 times the upper limit of the normal range (ULN), including alanine aminotransferase (ALT), aspartate aminotransferase (AST), or alkaline phosphatase (ALP).
9. Impaired renal function as determined by the Investigator, based on an estimated glomerular filtration rate (eGFR) < 90mL/min/1.73 m2 at Screening.
10. Pregnant or lactating at Screening or planning to become pregnant (self or partner) at any time during the study, including up to 30 days after study drug administration (for female participants) or up to 90 days after study drug administration (for female partners of male participants).
11. Fever or symptomatic viral or bacterial infection at time of Screening. Testing for SARS-CoV-2 infection will be performed in accordance with local guidelines (health authorities, Institutional Review Boards/Independent Ethics Committees, and study centre policies) and at the discretion of the Investigator, if required.
12. Participants who have received live vaccines or attenuated vaccines within 1 month before dosing. Participants may receive vaccination for SARS-CoV-2 at the discretion of the Investigator as soon as they are eligible, and a vaccine is available.
13. The participant has, according to World Health Organization (WHO) Grading, a cortical cataract greater than one-quarter of the lens circumference (Grade cortical cataract-2 [COR-2]) or a posterior subcapsular cataract > 2mm (Grade posterior subcapsular cataract-2 [PSC-2]). Participants with nuclear cataracts will not be excluded.
14. The participant is currently receiving, or has received within the past month, potentially cataractogenic medications, including a chronic regimen (more frequently than every 2 weeks) of any route of corticosteroids (limited to medium and high-potency topical steroids; intranasal steroids are acceptable) or any medication that may cause cataract (such as phenothiazines and miotics, amiodarone, allopurinol, and phenytoin), according to the Prescribing Information.
15. Positive test for hepatitis C antibody (HCV), hepatitis B surface antigen (HBsAg), or human immunodeficiency virus (HIV) antibody at Screening.
16. Participants with a positive toxicology screening panel (urine test including qualitative identification of barbiturates, tetrahydrocannabinol (THC), amphetamines, benzodiazepines, opiates and cocaine), or alcohol breath test.
17. Participants with a history of substance abuse or dependency or history of recreational intravenous (IV) drug use over the last 5 years (by self-declaration)
18. Regular alcohol consumption defined as >21 alcohol units per week (where 1 unit = 284mL of beer, 25mL of 40% spirit, or a 125mL glass of wine). Participant is unwilling to abstain from alcohol beginning 48 hours prior to admission to the CRU until completion of the primary Follow-up visit. (Part A [except Cohort A3]: Day 7; Part A [Cohort A3]: Day 35; Part B: Day 21).
19. Use of any IP or investigational medical device within 30 days prior to Screening, or 5 half-lives of the product (whichever is the longest) or participation in more than four investigational drug studies within 1 year prior to screening.
20. Use of any prescription medications (other than hormonal contraception: OCPs, long-acting implantable hormones, injectable hormones, a vaginal ring or an IUD), over the-counter (OTC) medication, herbal remedies, supplements or vitamins 2 weeks prior to dosing and during the course of the study without prior approval of the Investigator and MM. Simple analgesia (paracetamol, nonsteroidal anti-inflammatory drug [NSAID]) may be permitted at the discretion of the Investigator.
21. History of anaphylaxis or other severe allergy to any drug, food, toxin, or other exposure.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2021-06-08 (Actual); Primary Completion 2022-06-20 (Actual); Study Completion 2022-06-20 (Actual)

PRIMARY OUTCOMES:
To assess the safety and tolerability measures of AL01211 through Adverse Events/Serious Adverse Events in healthy adult participants | Baseline to End of the Treatment assessed up to an average of 90 days
  Number of participants with treatment related adverse events as assessed through CTCAE v5.0

SECONDARY OUTCOMES:
To assess the pharmacokinetics of AL01211 in healthy adult participants | Baseline to End of the Treatment assessed up to an average of 56 days
  The following parameters are used for pharmacokinetics: AUC0-last, AUC0-24h
Measurement of glucosylceramide in plasma and urine following oral dosing of AL01211 | Baseline to End of the Treatment assessed up to an average of 56 days
  Change in glucosylceramide levels
Measurement of monosialodihexosylganglioside in plasma and urine following oral dosing of AL01211 | Baseline to End of the Treatment assessed up to an average of 56 days
  Change in monosialodihexosylganglioside levels

CONTACTS AND LOCATIONS:
Overall Officials: Philip Ryan, MBBS, FRACP, Principal Investigator — Nucleus Network Pty Ltd.
Locations (1):
- Nucleus Network, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No